CLINICAL TRIAL: NCT05925322
Title: Brain Changes During Social Reward Psychotherapy for Mid- and Late-Life Suicidality: A Precision Imaging Trial
Brief Title: Brain Changes During Social Reward Psychotherapy for Mid- and Late-Life Suicidality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-05026093; R01MH133953 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-06-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Depression; Suicidal Ideation; Major Depressive Disorder; Depressive Disorder
Keywords: Late Life Depression; Psychotherapy; Mechanisms of Action; Positive Valence System; Social Reward
MeSH Terms: conditions — Depression; Suicidal Ideation; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Engage & Connect" Psychotherapy (Experimental): Engage & Connect is a remotely-delivered psychotherapy, aimed to increase engagement in rewarding social activities and in turn, reduce suicidality. In Engage & Connect, depressed middle-aged and older adults with suicidal ideation work with a therapist to develop "action plans" to pursue rewarding social activities of their choice.
  Interventions: Behavioral: "Engage & Connect" Psychotherapy
- Symptom Review and Psychoeducation (SRP) (Active Comparator): In this intervention, the therapist will review the participant's symptoms and provide literature-based clinical explanations and clarifications about the symptoms, the course, and the causes of depression and aging processes. In SRP, the therapist reviews the depressed individual's symptoms, and level of information on depression, identifies misconceptions, and guides selection of educational material which could benefit the patient.
  Interventions: Behavioral: Symptom Review and Psychoeducation (SRP)

INTERVENTIONS:
Behavioral: "Engage & Connect" Psychotherapy — 9-weeks of weekly psychotherapy sessions focused on social reward exposure
  Arms: "Engage & Connect" Psychotherapy
Behavioral: Symptom Review and Psychoeducation (SRP) — 9-weeks of weekly psychotherapy sessions focused on symptom review and psychoeducation about depression and aging
  Arms: Symptom Review and Psychoeducation (SRP)

SUMMARY:
The investigators hypothesized that during the 9-week course of Engage & Connect treatment there will be an increase in brain functions of the Positive Valence System which in turn will lead to reduction in suicidality.

DETAILED DESCRIPTION:
Social disconnection peaks in middle and late life and leads to an increased risk of suicide, persistent depression, and poor response to psychosocial interventions. There is a critical need to develop a mechanistic understanding of the link between social disconnection and suicidality, identify biological targets, and address targets with scalable interventions. The investigators developed a novel psychotherapy, Engage & Connect, aimed to improve functions of the Positive Valence System (PVS) that are impaired in suicidality through increased engagement in rewarding social activities. This study will use state-of-the-art precision imaging methods and clinical measures to evaluate brain- and behavioral changes in the PVS during psychotherapy.

Participants will:

* Be randomly assigned to 9-weekly sessions of either Engage & Connect therapy or Symptom Review and Psychoeducation
* Complete 4 research assessments
* Complete 3 MRI scans

ELIGIBILITY:
Inclusion Criteria:

* Ages aged 50-80 [stratified so that 50% are older than 65]
* Endorsement of Suicidal Ideation [Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders-5 (SCID-5) Suicide Item (Item 9) with a score of 2
* Major Depressive Disorder as determined by the SCID-5
* Depression Rating Scale [Montgomery-Åsberg Depression Rating Scale (MADRS)] score of 16 or greater.
* Mini Mental Status Exam (MMSE) equal or greater than a score of 23
* Off antidepressants or on a stable dose of an antidepressant for 8 weeks and do not intend to change the dose in the next 10 weeks, without individual psychotherapy services during the study period.
* Capacity to provide consent for research assessment and treatment.

Exclusion Criteria:

* Intent or plan to attempt suicide in the near future.
* History or presence of psychiatric diagnoses other than major depressive disorder without psychotic features, generalized anxiety disorder, or specific phobia.
* Use of psychotropic drugs or cholinesterase inhibitors other than use of 0.5 mg or less of lorazepam daily up to seven times per week.
* Neurological disorders (dementias, amnestic and multidomain Mild Cognitive Impairment, Parkinson's disease, epilepsy, etc.).
* Acute or severe medical illness in the past 3 months (metastatic cancer, multiple sclerosis, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction, cardiac, renal, or respiratory failure; severe chronic obstructive pulmonary disease, etc.) that may be the primary cause depressive symptoms, influence brain systems of interest, or impact ability to participate in the study.
* Contraindications to MRI scanning including cardiac pacemaker, heart valve replacement, vascular stent, insulin pump, cochlear implant, any other metallic biomedical implant contraindicating to MRI, and claustrophobia.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in resting state functional connectivity of the Positive Valence System | Baseline, midtreatment (week 6) and post treatment (week 9)
  Change in resting state fMRI connectivity of functional networks representing structures previously associated with the Positive Valence System (Dorsal anterior cingulate cortex [dACC], the Subgenual Anterior Cingulate Cortex [sgACC], and the basal forebrain/nucleus accumbens [NAcc]). The investigators will also test between-network connectivity between the positive valence system and the default mode-, salience-, and fronto-parietal networks. Functional connectivity within- and between-network will be measured with a correlational score of 0 to 1, with 0 being the lowest and 1 being the highest.
Change in STAR task reaction time following social feedback | Baseline, midtreatment (week 6), and post treatment (week 9)
  "The Social Task for Assessment of Reward" is a computerized task that measures response to social rewards. Reaction time will be measures in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Nili Solomonov, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after de-identification, as well as study protocol, treatment manuals, statistical analysis plan and informed consent. The investigators will also share the fMRI tasks and analytic code by request with all interested researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the investigators publish the main results, they will make de-identified data available to other researchers, under a data-sharing agreement overseen by the DSMB, and in compliance with policy of the IRB and NIMH.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. All researchers requesting data will commit to using the data solely for research purpose; secure the data; return or destroy it once analyses are completed; do not share it with other researchers.